CLINICAL TRIAL: NCT03364647
Title: The Effect of Various Strength Training Protocols in ACL Reconstructed Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brian W. Noehren (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Brian W. Noehren, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-0750-F6A; R01AR071398 (NIH)
Record Dates: First submitted 2017-11-15; First posted 2017-12-06 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear; Physical Therapy
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, outcomes assessors, and the PI will be blinded as to the participant's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Blood flow restriction training (Experimental): Group will use blood flow restriction training and standard of care
  Interventions: Other: Arm A - blood flow restriction training
- Arm B - standard of care plus sham (Sham Comparator): Group will receive standard of care plus a sham version of blood flow restriction training
  Interventions: Other: Arm B - standard of care

INTERVENTIONS:
Other: Arm A - blood flow restriction training — Group receive standard of care plus blood flow restriction training
  Arms: Arm A - Blood flow restriction training
Other: Arm B - standard of care — Group will receive standard of care plus a sham version of blood flow restriction training
  Arms: Arm B - standard of care plus sham

SUMMARY:
The purpose of the study is to determine how two different blood flow restriction training programs used in conjunction with standard rehabilitation affect leg strength. By doing this study, the investigator hopes to learn if one program improves strength and function more than the other. The investigator also hope to learn how the training affects the properties of muscle in participants who will or have had anterior cruciate ligament (ACL) reconstruction. These results will help define how the training programs are working.

There will be no charge to the participant for their physical therapy visits as long as they are part of the study

The initial visit and follow up assessment at the end of the training will each take up to 6 hours (2 hours for MRI, 2 muscle biopsy, 2 for muscle strength, movement mechanics and questionaires).

The physical therapy visits will range from 60-120 minutes depending on the participant's stage of recovery and the activities to engage in. Training sessions will be held 3 days a week for approximately 4 weeks before surgery and up to 24 weeks after surgery. There will be a total of 4 additional study visits over a 7 month period. The first visit will be used to capture baseline conditions of their knee and thigh muscles (muscle biopsy, MRI, strength). The second visit will occur right before surgery to assess changes during prehabilitation (strength and walking mechanics). The third visit will occur 4-5 months after surgery and will be a complete reevaluation of their thigh muscle and knee function (muscle biopsy, MRI, strength, gait). The last visit will occur 6-7 months after surgery and will involve an assessment of their thigh muscle strength, walking, and jumping form.

The muscle biopsy and magnetic resonance imaging portion of the study will occur in the outpatient unit of the Center for Clinical and Translational Science at the UK Medical Center and the MRI center located on the medical center campus. The muscle biopsy will take an additional 15 minutes and the MRI up to two hours (1 hour per leg). It can take up to 4 hours total to complete both procedures. The investigator will accommodate participant preference for scheduling.

DETAILED DESCRIPTION:
The following procedures may be performed.

Training sessions: Participants will be randomly assigned one of two groups. Assignments to which group are determined by random assignment based upon participant's number. One group will receive standard of care and the other will receive standard of care plus blood flow restriction training.

The air bands will then be placed on the participant's thighs and they will be doing a standardized exercise program that will vary depending on the stage of rehabilitation they are in and as determined by the study personnel. Participants will also complete a standardized course of physical therapy. Activities in physical therapy may include ice over the knee, range of motion exercises to maintain hip strength and gait training exercises as needed and as the participant's impairments dictate. The investigator will also provide an educational program at regular intervals on the injury and recovery.

Quadriceps strength: Participants will sit in a seated position and a stabilizing strap will be placed around the thigh. A second strap will be placed around the bottom of their lower leg and attached to the isokinetic dynamometer (a muscle strength testing device) which will control movements and apply force at several different speeds and in a isometric mode.

Motion Analysis: Motion analysis will provide a means for evaluating motion of the participant's hip, knee and ankle joints during walking and jogging on the treadmill. Participants will have reflective markers placed on certain landmarks of their legs and lower back to allow the motion analysis system to record their trunk, hip, knee, and ankle movements. Markers will be applied with sticky tape to the skin and if necessary, athletic tape to limit marker movement during activities. A stationary trial will be collected to help the researcher identify anatomical landmarks. Motion data will be collected for 10 seconds every minute. Participants will perform a series of jumps on both legs and on a single leg. In addition participants will be asked to go up and down step.

Treadmill Activity: Participants may walk on the treadmill as long as necessary to feel comfortable with it. Once ready, participants will walk at a self-selected warm up pace for 5 minutes. The investigator will then gradually increase the speed 1.5 m/s for 2 minutes each. The speed of the treadmill will then be increased gradually to a self-selected comfortable jogging\running pace for 2 minutes. Participants may request to stop at any time.

Muscle Biopsy: A small piece of muscle tissue will be removed from both of thighs. The muscle tissue will be taken from the outside of your thigh and will be taken about one hand width above your knee. A 1 inch by 1 inch portion of hair will possibly need to be shaved if necessary. The area of thigh will be numbed and a small ¼ inch incision will be made in the skin. A needle will then be briefly (lasting just a couple of seconds) inserted into the muscle to remove a .005 ounce piece of muscle (about the size of a pencil eraser). The incision will be pulled closed with a band-aid after the site is cleaned with an alcohol preparation and the participant's leg will be wrapped snugly with an elastic bandage. The procedure will last approximately 15 minutes. The tissue samples will be used in the analysis process. In addition, standard venipuncture methods will be used to collect one 7.5 mL tube of blood to be used for analysis.

Magnetic Resonance Imaging & Spectroscopy Center: Participants will be asked to complete a medical screening questionnaire that will ask specific questions about their health and medical history. This information will be used to determine eligibility to participate in the study. At this time, the procedures and risks involved in participating in the research study will be explained to the individual. Participants will also fill out a questionnaire asking whether they have any metal in their body as well as any other medical conditions that may need to be considered before they enter the MRI scanner. The metal screening questionnaire will be reviewed by the individual operating the scanner and if any risks are identified, the participant may not be able to participate.

Participants will be taken to the MRI scanner by the experimenter. Participants will be asked to remove all jewelry, body piercings, hair accessories, belts, wallets, credit cards, and loose change and leave these items with the experimenter. Participants will then be instructed about specific MRI procedures.

The magnetic resonance scanning will take approximately 60 minutes per leg. Participants will be asked to lie still during the scanning.

ELIGIBILITY:
Inclusion Criteria:

* ACL tear and no previous ACL reconstruction on either the involved or other limb

Exclusion Criteria:

* Previous surgeries or conditions that might affect gait
* Any current condition other than ACL or meniscus injury which might affect gait
* Unable to provided informed consent
* Diabetic or have uncontrolled hypertension
* Have recent inflammation, bleeding disorders, active bleeding or infection within the lower limbs.
* Allergic to Betadine or Xylocaine HCL.
* Taking warfarin/Coumadin, clopidogrel/Plavix, Rivaroxaban/Xarelto, Dabigatran/Pradaxa that may cause excess bleeding.
* Any implanted medical device
* A history of deep vein thrombosis, have a family history of deep vein thrombosis, or varicose veins
* Spinal fusion
* Inability able to attend regular physical therapy or study visits
* Injury occurring more than ten weeks prior to study enrollment
* Not skeletally mature (growth plates not closed)

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Noehren, PT., Ph.D, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky Orthopaedics and Sports Medicine Center, Lexington, Kentucky
  - University of Kentucky BioMotion Laboratory, 725 Rose Street, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erickson LN, Owen MK, Casadonte KR, Janatova T, Lucas K, Spencer K, Brightwell BD, Graham MC, White MS, Thomas NT, Latham CM, Jacobs CA, Conley CE, Thompson KL, Johnson DL, Hardy PA, Fry CS, Noehren B. The Efficacy of Blood Flow Restriction Training to Improve Quadriceps Muscle Function after Anterior Cruciate Ligament Reconstruction. Med Sci Sports Exerc. 2025 Feb 1;57(2):227-237. doi: 10.1249/MSS.0000000000003573. Epub 2024 Oct 1. PMID 39350350
- [Derived] Erickson LN, Lucas KCH, Davis KA, Jacobs CA, Thompson KL, Hardy PA, Andersen AH, Fry CS, Noehren BW. Effect of Blood Flow Restriction Training on Quadriceps Muscle Strength, Morphology, Physiology, and Knee Biomechanics Before and After Anterior Cruciate Ligament Reconstruction: Protocol for a Randomized Clinical Trial. Phys Ther. 2019 Aug 1;99(8):1010-1019. doi: 10.1093/ptj/pzz062. PMID 30951598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Department of Orthopaedic Surgery & Sports Medicine at the University of Kentucky and were scheduled to undergo surgical reconstruction by one of three orthopedic surgeons.
Pre-assignment Details: 647 participants were assessed for eligibility. Of those, 592 participants were excluded due to not meeting inclusion criteria or declining to participate. 55 participants were randomized of which 26 received the allocated intervention (BFRT) and 26 received the SHAM intervention. 3 participants withdrew after being randomized but before receiving the intervention.
Period: Overall Study
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
Started | 26 | 26
Completed | 23 | 25
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (6.0) | 21.2 (5.3) | 21.0 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 15 | 15 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.3 (4.2) | 25.7 (4.4) | 25.4 (4.5)
Time since injury [Mean (Standard Deviation); unit: Days] | 20.2 (16.5) | 24.3 (16.7) | 22.3 (16.9)
Graft Type [Count of Participants; unit: Participants]
  Patellar | 24 | 24 | 48
  Hamstring | 1 | 2 | 3
  Unknown (lost to follow up before surgery) | 1 | 0 | 1
Meniscal Injury [Count of Participants; unit: Participants]
  Lateral | 1 | 4 | 5
  Medial | 7 | 6 | 13
  Both | 16 | 14 | 30
  None | 1 | 2 | 3
  Unknown (lost to follow up before surgery) | 1 | 0 | 1
Weight Bearing Status After Surgery [Count of Participants; unit: Participants]
  Weight Bearing as Tolerated | 23 | 25 | 48
  Non-weight Bearing | 2 | 1 | 3
  Unknown (lost to follow up before surgery) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Measure Change in Isometric Peak Torque Quadriceps Strength
Description: Assessed with a Biodex Multi-Joint System 4 Isokinetic Dynamometer. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Time Frame: Baseline, and post-surgery (up to 5 months)
Measure: Mean (Standard Deviation); unit: Nm/Kg
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
Number analyzed (Participants) | 23 | 25
Nm/Kg
  Baseline | 2.18 (0.66) | 2.06 (0.65)
  Post-surgery | 1.96 (0.59) | 1.95 (0.57)

2. Primary Outcome: Measure Change in Isokinetic Peak Torque Quadriceps Strength
Description: as for outcome 1
Time Frame: Baseline and post-surgery (up to 5 months)
Population: 1 participant excluded from isokinetic strength measurement due to injury
Measure: Mean (Standard Deviation); unit: Nm/kg
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
Number analyzed (Participants) | 22 | 25
Nm/kg
  Baseline | 1.03 (0.35) | 1.00 (0.41)
  Post-surgery | 1.13 (0.33) | 1.09 (0.38)

3. Primary Outcome: Measure Change in Rate of Torque Development
Description: Isokinetic Dynamometer will be used. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Time Frame: Baseline and post-surgery (up to 5 months)
Measure: Mean (Standard Deviation); unit: Nm/kg/s
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
Number analyzed (Participants) | 23 | 25
Nm/kg/s
  Baseline | 7.10 (3.46) | 6.35 (3.14)
  Post-surgery | 5.51 (2.79) | 4.68 (2.37)

4. Secondary Outcome: Measure Change in Quadriceps Muscle Morphology - T1Rho Relaxation Time
Description: MRI will be used. Analyses may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Time Frame: Baseline, Post-surgery (up to 5 months)
Population: Participants included in MRI analysis
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
Number analyzed (Participants) | 20 | 20
milliseconds
  Baseline | 0.029 (0.003) | 0.031 (0.004)
  Post-surgery | 0.030 (0.002) | 0.029 (0.002)

5. Secondary Outcome: Measure Change in Quadriceps Muscle Morphology - Physiological Cross-sectional Area (PCSA)
Description: as for outcome 4
Time Frame: Baseline, Post-surgery (up to 5 months)
Population: Participants included in MRI analysis for this measure
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
Number analyzed (Participants) | 18 | 19
mm2
  Baseline | 6238.7 (1783.0) | 6290.9 (1942.5)
  Post-surgery | 6626.0 (2484.6) | 6386.6 (1862.2)

6. Secondary Outcome: Measure Change in Knee Biomechanics - Peak Knee Flexion
Description: 3D Motion Capture will be used. The primary analysis may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Time Frame: Baseline and post-surgery (up to 5 months)
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
Number analyzed (Participants) | 23 | 25
degrees
  Baseline | 21.51 (4.66) | 22.50 (4.42)
  Post-surgery | 16.87 (8.05) | 16.63 (4.76)

7. Other Pre Specified Outcome: Measure the Change in Muscle Physiology After Using BFRT for Treatment in Patients Who Will Have an ACL Reconstruction.
Description: Muscle biopsy, which may include immunohistochemistry, histochemistry, protein expression, gene expression, or single fiber morphology may be measured. Analyses may include the comparison of these observations over multiple time points, with a particular interest in whether there are between-group or within-patient differences.
Time Frame: Before surgery, 4 months after surgery
Reporting Status: Not Posted

8. Secondary Outcome: Measure Change in Knee Biomechanics - Knee Extensor Moment (KEM)
Description: as for outcome 6
Time Frame: Baseline and post-surgery (up to 5 months)
Measure: Mean (Standard Deviation); unit: (Nm/(kg*m)
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
Number analyzed (Participants) | 23 | 25
(Nm/(kg*m)
  Baseline | 0.16 (0.11) | 0.19 (0.12)
  Post-surgery | 0.16 (0.16) | 0.13 (0.14)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Arm A - Blood Flow Restriction Training | Arm B - Standard of Care Plus Sham
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Blood Flow Restriction Training (N=23) | Arm B - Standard of Care Plus Sham (N=25)
Patellar Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03364647/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT03364647/ICF_000.pdf